CLINICAL TRIAL: NCT07167043
Title: Reasoning Artificial Intelligence Collaborate With Radiologists in Neurological Disease Interpretation and Diagnosis on CT and MRI
Brief Title: An Explainable Neuroradiologist Artificial Intelligence Assistance System for Brain CT and MRI
Status: Enrolling by invitation | Type: Observational
Sponsor: Yaou Liu (Other)
Responsible Party: Sponsor-Investigator, Yaou Liu, Director of the Radiology Department, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Other Study IDs: 2025-A09
Record Dates: First submitted 2025-09-03; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Central Nervous System Disease; MRI; CT; AI (Artificial Intelligence); Radiology
MeSH Terms: conditions — Central Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Biospecimen is not stored beyond the timeframe of this study, for the purpose of this study. However, biospecimen is stored beyond the timeframe of this study, for the purpose of regular clinical care. In this case, biospecimen refers to histopathology tissue acquired from confirmatory brain biopsies. Within the scope of clinical routine, storing such specimen can facilitate reassessments through the future, e.g. for comparisons if the patient presents new findings or metastasis of their initial findings, for comparisons against histopathology findings of the original patient's offspring, or even for legal purposes in the case of misdiagnosis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: AI-assisted diagnostic systems — Diagnosing neurological diseases on CT/MRI with and without AI-assisted tools

SUMMARY:
This clinic trial aims to validate the working performance of radiologists with or without artificial intelligence (AI) diagnostic tool at neurological diseases diagnosis on brain CT/MRI. Routine diagnosis workflow in real clinical scenario including imaging reading, feature interpretation, differential diagnosis, writing initial report and optimizing revised version. And the gold standards of diagnosis are the histopathology references for brain tumors and the discharge diagnosis integrating all the examination results for the other neurological diseases. The performance of AI-assisted tools on diagnosing should be examined in a clinical process with multiple aspects identical to human radiologists' work before being transformed and putted to use. This study hypothesizes that AI models, trained with over 100,000 patient scans, are non-inferior to radiologists in neurological disease diagnosis on brain CT and MRI. For the secondary end-points, we investigate the performance of AI-radiologist collaboration of reasoning-enhanced AI-assisted systems. We hypothesize that, by visualizing the process of imaging interpretation and diagnosis, reasoning-enhanced AI can not only improve working performance of radiologists but also boost their trust in AI tools.

DETAILED DESCRIPTION:
Neurological diseases affect over 50% of the world population, which contribute to an increasingly needs of imaging examination for screening and diagnosis. The shortage of neuroradiologists led to the excessive workload, linked with increasing of error rates and decreasing of report quality. Inexperienced radiologists struggle to make accurate diagnoses for some neurological diseases, especially brain tumors, which may lead to additional delays and a potentially meaningless examination for patients.

Artificial intelligence (AI) has shown potential to be "a tireless resident", which can rival human performance in medical imaging interpretation and assist radiologists in multiple links of clinical diagnostic work. However, clinicians recognize that "Black-box" models lacking clinical utility and interpretability face significant barriers to real-world deployment. While the reasoning-enhanced AI model, trained by a hundred thousand data, can not only achieve accurate and efficient diagnosis but also but also address the lack of explainability, transparency, and trust.

Owing to the heterogeneity of multi-modal real clinical data and complexity of neurological diseases, whether the developed AI-assisted system can truly serve as an "AI resident" facing challenges and doubts. Clinical trial is the best approach to verify the performance of diagnosis and human-machine collaboration of AI model with a wide range of users and prospective data before being approved for clinical use. Key aspects of the study design have been established in conjunction with a multi-disciplinary scientific advisory board, consisting with experts in AI, radiology, neurology, and pathology, to ensure meaningful validation of reasoning-enhanced AI model towards clinical translation.

This clinic trial contains two sub-studies:

1. Clinical silence trial study for AI tools only:

   There are three approaches may be used in this stage to compare the working performance of our AI model with radiologists and the other models.

   First, a curated mini-dataset of totally 1,000 scans of brain tumor cases on MRI and cerebrovascular disease cases on brain CT will be publicly released. Teams can use this dataset to train or test on their AI models, and submit their trained algorithms or prediction results for evaluation. The performance of the uploaded models will be tested on the same testing cohort of us, and the uploaded prediction results will be compared with the generated content of us.

   Second, a fine-tuned offline AI-assisted systems will be embedded in the picture archiving and communication system (PACS) in the radiology department after getting permission of medical affairs department and ethics committee in some medical centers. However, radiologists in these medical centers will not get AI-generated diagnoses and reports during this stage, while the imaging reports of brain MRI and CT generated by AI and radiologists will be recorded at the same time.

   Third, prospective data of brain MRI and CT with corresponding imaging reports and gold standard diagnostic results will be collected from all over the world as the test data inputting to our AI model.

   Finally, the consistency and accuracy of the report between AI models and radiologists will be compared, with respect to the histopathology and discharge diagnosis (< 3 month) as reference.
2. AI-radiologist collaboration study:

In this stage, we aim to perform generalization verification on our reasoning-enhanced neuroimaging AI in the real clinical scenarios.

Over 50 international radiologists will be recruited to perform a diagnosis study using a subset of 400 scans from the testing cohort of us. The workflow including such steps in order: imaging reading, writing initial report, making diagnosis, reading AI reasoning, revising initial report, and evaluating content generated by AI. When writing reports, radiologists will be will be randomly assigned to two groups and asked to complete half of cases with AI-assisted tools and the other half of cases without, to ensure every case will be completing by two radiologists of the same level with and without AI assistance, respectively.

The first goal of this study is to estimate the performance of the average radiologist with or without AI as well as their working efficiency and confidence at neurological diseases diagnosis on CT and MRI.

The secondary goal is to evaluate the clinical viability and superiority of reasoning-enhanced AI on human-machine collaborative task. The accuracy and completion will be compared between revised reports with initial version written by radiologists, while radiologists' inclination and diagnostic confidence will be recorded as subjective evaluation indexes.

ELIGIBILITY:
Inclusion Criteria:

* For MRI: patients suspected of harboring brain tumors or detected with brain occupancy at initiating or other institution, who subsequently underwent brain MRI.
* For CT: patients with or without neurological symptoms, suspected of harboring ischemic, hemorrhagic, space-occupiing, degenerative brain disease, or traumatic brain injury, who subsequently underwent brain CT.

Exclusion Criteria:

* Patients who opted-out or did not give permission to reuse clinical data.
* Patients with a history of prior brain surgery.
* Patients whose brain CT or MRI exhibit severe artifacts (e.g. heavy warping due to air, metal artifacts, heavy motion artifacts), thereby impeding the usage of the data.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patient exams are of men suspected of harboring brain tumors or the other neurological diseases, with or without neurological symptoms, and without a history of prior brain surgery. Patients underwent brain CT and MRI, and were primarily examined at Beijing Tiantan hospital, between 2012-2026.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
AI tools vs Radiologists from Clinical silence trial | 6 months
  Diagnostic performance of AI models and over 50 radiologists from the Clinical silence trial study, at neurological diseases on brain CT/MRI, with respect to histopathology and discharge diagnosis as reference, to assess the working performance of neuroimaging AI diagnostic tools.
AI-assisted diagnostic tool collaborates with Radiologists in clinical workflow | 6 months
  Working efficiency (time taking) and diagnostic confidence and accuracy of radiologists from AI-radiologist collaboration study, at neurological diseases on brain CT/MRI, to assess the clinical viability of AI-assisted diagnostic tool.

SECONDARY OUTCOMES:
Present AI vs the other AI tools uploaded from Clinical silence trial | 6 months
  Diagnostic performance of our AI models and the others uploaded from Clinical silence trial, at neurological diseases on brain CT/MRI, with respect to histopathology and discharge diagnosis as reference, to deduce the optimal AI models in diagnosis and report generation of neurological diseases.
Reasoning-enhanced AI model collaborates with Radiologists in clinical workflow | 6 months
  Diagnostic confidence and accuracy of radiologists from AI-radiologist collaboration study, at neurological diseases on brain CT/MRI, and their trust in AI, to assess the value and clinical viability of AI model with visualized reasoning process.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, China